CLINICAL TRIAL: NCT04939649
Title: Ketamine As an Adjunctive Therapy for Major Depression - a Randomised Controlled Trial: [KARMA-Dep (2)]
Brief Title: Ketamine As an Adjunctive Therapy for Major Depression (2)
Acronym: KARMA-Dep2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Prof Declan McLoughlin, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRFSPN004; 2019-003109-92 (EudraCT Number)
Record Dates: First submitted 2021-06-20; First posted 2021-06-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Episode; Unipolar Depression; Bipolar Depression
Keywords: ketamine; glutamate
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participants will receive up to a four-week course of twice-weekly infusions of ketamine at 0.05mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Participants will receive up to a four-week course of twice-weekly infusions of midazolam at 0.045mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — A sub-anaesthetic dose of ketamine will be administered for up to a four-week course of twice-weekly infusions.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — A sub-anaesthetic dose of midazolam will be administered for up to a four-week course of twice-weekly infusions.
  Other Names: Hypnovel
  Arms: Midazolam

SUMMARY:
Pragmatic, randomised, controlled, parallel-group, superiority trial of ketamine vs. midazolam as an adjunctive therapy for depression. The main purpose of the trial is to assess the mood-rating score difference between ketamine and midazolam from before the first infusion to 24 hours after the final infusion, supplemented by a 95% confidence interval. There will also be a 24-week follow-up after the final infusion session.

DETAILED DESCRIPTION:
Pragmatic, randomised, controlled, parallel-group, superiority trial. Trial participants will be patients admitted to St Patrick's University Hospital for treatment of a major depressive episode. The investigators aim to recruit up to 104 participants who will be eligible for this study and randomly allocate 52 patients to each group. Both participants and assessors will be blind to treatment allocation. Eligible consented participants will be randomly allocated in a 1:1 ratio to a course of up to eight infusions of either ketamine or midazolam twice weekly over up to four weeks. Block randomisation will be independently performed. Physical, psychotomimetic and cognitive outcomes will be monitored before, during and after infusions. During the allocated infusions and follow-up period patients will be monitored for treatment-related adverse events relating to both mental and physical health. Participants will also be followed-up for 24 weeks after the end of the initial randomised treatment and assessment period lasting up to four weeks, in order to identify if and when relapse occurs. During the trial, both groups will continue usual inpatient care as prescribed by their treating team.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Montgomery-Åsberg Depression Rating Scale (MADRS) score ≥ 20 at screening and start of the first infusion.
* Voluntary admission for treatment of an acute depressive episode
* Meet DSM-5 criteria for a major depressive disorder or bipolar affective disorder (current episode depression). Diagnosis of a major depressive disorder or bipolar affective disorder (DSM-5) will be confirmed by the structured diagnostic Mini International Neuropsychiatric Interview (MINI; updated Version 7 for DSM-5).

Exclusion Criteria:

* Current involuntary admission.
* Medical condition rendering unfit for ketamine/midazolam.
* Currently taking any of the contraindicated medications that may alter the pharmacokinetics of ketamine.
* Active suicidal intention.
* Dementia.
* Lifetime history of schizophrenia or schizoaffective disorder; active anorexia nervosa or bulimia nervosa in the past 12 months; alcohol or other substance use disorder (with the exception of nicotine) in the previous six months; any DSM-5 disorder other than a major depressive episode (unipolar or bipolar) as the primary presenting problem.
* Electroconvulsive Therapy (ECT) administered within the last two months.
* Pregnancy, breastfeeding or considering becoming pregnancy whilst on the trial for up to 12 weeks after last dose or inability to confirm use of adequate contraception during the trial.
* Breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale-10 item version (MADRS) | 28 weeks
  The MADRS is a validated, 10-item, observer-rated scale that measures the symptoms and severity of depression. The primary outcome measure will be the change from baseline in the MADRS score to 24 hours after the final infusion.
  MADRS will be completed at screening (prior to randomisation), before and after all infusion sessions (at the following timepoints: -40 (±20) mins before the infusion begins; +60 (±10) mins and +120 (±10) mins after the infusion begins; +24 (±1) hours after the infusion ends) and at the 6, 12 and 24 weeks follow-up time points. Sleep and appetite scores will be carried over from -40 minutes to +60 minutes, +120 minutes, and 24 hours after each infusion.
  Response to treatment is defined as a ≥50% improvement from baseline MADRS score. Remission is defined as achieving a MADRS score ≤10. For those deemed to be treatment remitters, relapse at follow-up time points is defined as a MADRS score of ≥18.

SECONDARY OUTCOMES:
The Clinician-Administered Dissociative States Scale (CADSS) | 4 weeks
  The CADSS will measure dissociative symptoms, as a possible subjective side effect of either ketamine or midazolam. The CADSS consists of 23 items and scores for each item range from 0 to 4. The CADSS measures dissociative symptoms in the following domains: identity, proprioception, time perception, colour and depth perception, and other modalities. The maximum score is 92, with higher scores indicating more dissociative symptoms.
  The CADSS will be completed three times at each infusion session: before (-30 (±10) mins before the infusion begins), during (+30 (±5) mins after the infusion begins) and after (+60 (±10) mins after the infusion begins, i.e. 20 (±10) mins after the infusion ends).
The Brief Psychiatric Rating Scale (BPRS) | 4 weeks
  The positive symptoms subscale of the BPRS will be used to measure psychotomimetic effects of either ketamine or midazolam. This 4-item positive symptoms subscale measures suspiciousness, hallucinations, unusual thought content, and conceptual disorganisation. Each item is scored between 0 and 7. The maximum score is 28, with higher scores indicating more severe psychotic symptom.
  Participants will complete the BPRS three times at each infusion session: before (-30 (±10) mins before the infusion begins), during (+30 (±5) mins after the infusion begins) and after (+60 (±10) mins after the infusion begins, i.e. 20 (±10) mins after the infusion ends).
Young Mania Rating Scale (YMRS; mood item) | 4 week
  The YMRS is an observer-rated assessment tool for severity of mania and hypomania. The single mood item of the YMRS, rated from 0 to 4 (representing a range from normal mood to frank euphoria), will be used to assess for possible mood elevation during the infusion sessions. Higher scores reflect more elevated mood.
  Participants will have the YMRS performed three times at each infusion session: before (-30 (±10) mins before the infusion begins), during (+30 (±5) mins after the infusion begins) and after (+60 (±10) mins after the infusion begins, i.e. 20 (±10) mins after the infusion ends).
Observer's Assessment of Alertness/Sedation; responsiveness subscale (OAA/S-R) | 4 weeks
  The OAA/S-R is an observer-rated assessment that will be used to measure levels of sedation experienced by participants during either ketamine or midazolam infusion. The OAA/S-R ranges in score from 1 to 5, where 1 denotes deep sleep (i.e. no response to mild prodding or shaking) and 5 denotes fully alert.
  The OAA/S-R will be completed three times at each infusion session: before (-30 (±10) mins before the infusion begins), during (+30 (±5) mins after the infusion begins) and after (+60 (±10) mins after the infusion begins, i.e. 20 (±10) mins after the infusion ends).
20-item Physician Withdrawal Checklist (PWC-20) | 16 weeks
  The PWC-20 will be used to assess for potential withdrawal symptoms during and after completion of the allocated course of ketamine/midazolam infusions. The PWC-20 is a brief checklist and each item is rated from 0 (not present) to 3 (severe). PWC-20 scores range from 0 to 60, with higher scores indicating more withdrawal symptoms with greater severity.
  The PWC-20 will be completed at screening (prior to randomisation), 24 (±1) hours after the end of the fourth and final infusions, and the 6- and 12-week follow-up timepoints.
The Quick Inventory of Depressive Symptoms, self-report version (QIDS-SR) | 28 weeks
  The QIDS-SR is a validated, self-report measure of depressive symptoms. The QIDS-SR consists of 16 items, with each item rated on a scale from 0 to 3. Total scores range from 0 to 48, with higher scores reflecting greater burden of depressive symptoms.
  The QIDS-SR will be completed at screening (prior to randomisation), before and after all infusion sessions (at the following timepoints: -40 (±20) mins before the infusion begins; +60 (±10) mins and +120 (±10) mins after the infusion begins; +24 (±1) hours after the infusion ends) and at the 6, 12 and 24 weeks follow-up time points. Sleep and appetite items 1,2,3,4,6,7,8 & 9 on the QIDS-SR will be carried over from -40 minutes before each infusion to +60 minutes, +120 minutes & 24 hours after each infusion in line with the methodology of previous literature.
Patient-Rated Inventory of Side Effects (PRISE) | 28 weeks
  The PRISE is a 9-item, self-report measure that will document general adverse events experienced by patients during each infusion, by identifying and evaluating the tolerability of each adverse event. The PRISE assesses adverse events in the following symptom domains; Gastrointestinal, Heart, Skin, Nervous System, Eyes/Ears, Genital/Urinary, Sleep, Sexual Functioning, and Other. Each domain has multiple symptoms which can be endorsed. For each domain the patient rate whether or not the symptoms are tolerable or distressing.
  The PRISE will be completed at screening (prior to randomisation), after all infusion sessions (+120 (±10) mins after the infusion begins), and at the 6, 12 and 24 weeks follow-up time points.
The Montreal Cognitive Assessment (MoCA) | 28 weeks
  The MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses the following cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation. The maximum score is 30, with higher scores indicating better cognition.
  The MoCA will be completed at screening (prior to randomisation), at +120 (±10) mins after the infusion begins during the first and final infusion sessions, and at the 12 and 24 weeks follow-up time points.
EuroQol-5 dimensions-5 level scale for health status (EQ-5D-5L) | 28 weeks
  Health-related quality-of-life will be measured using the EQ-5D-5L. The EQ-5D-5L consists of the EQ-5D descriptive system, and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system includes the following five dimensions that assess an individual's self-rated health status: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated on a 5-point Likert scale. The digits related to each response to the five dimensions are combined into a 5-digit number, which describes the patient's health state.
  The EQ VAS includes a vertical visual analogue as a quantitative measure of subjectively rated health, with endpoints labelled as 'Best imaginable health status' and 'Worst imaginable health status'.
  The EQ-5D-5L will be administered at screening (prior to randomisation) and at the 6-, 12- and 24-week follow up time periods.
Client Service Receipt Inventory (CSRI) | 28 weeks
  The CSRI will calculate healthcare costs using the following data: sociodemographic information, usual living situation, employment status and income levels and the care services and supports used by participants. Currently prescribed medicines will also be recorded.
  Healthcare costs will be estimated using the CSRI at baseline and at the 6-, 12- and 24-week follow-up timepoints.
Adverse events (AE) and serious adverse events (SAE) review | 28 weeks
  AEs and SAEs will be reviewed at every visit. All AEs and SAEs will be reported and followed up until resolved or until final visit.
Concomitant Medication | 28 weeks
  All medications taken one month prior to participant screening will be recorded. At all other visits, concomitant medication taken since last visit will be documented. Adherence to prohibited/contraindicated medication requirements will be assessed and documented at each infusion visit.

CONTACTS AND LOCATIONS:
Overall Officials: Declan M McLoughlin, PhD, Principal Investigator — University of Dublin, Trinity College and St Patrick's Mental Health Services
Locations (1):
- St Patrick's Univeristy Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jelovac A, McCaffrey C, Terao M, Shanahan E, Whooley E, McDonagh K, McDonogh S, Loughran O, Shackleton E, Igoe A, Thompson S, Mohamed E, Nguyen D, O'Neill C, Walsh C, McLoughlin DM. Serial Ketamine Infusions as Adjunctive Therapy to Inpatient Care for Depression: The KARMA-Dep 2 Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1216-1224. doi: 10.1001/jamapsychiatry.2025.3019. PMID 41123905
- [Derived] Jelovac A, McCaffrey C, Terao M, Shanahan E, Mohamed E, Whooley E, McDonagh K, McDonogh S, Igoe A, Loughran O, Shackleton E, O'Neill C, McLoughlin DM. Study protocol for Ketamine as an adjunctive therapy for major depression (2): a randomised controlled trial (KARMA-Dep [2]). BMC Psychiatry. 2023 Nov 16;23(1):850. doi: 10.1186/s12888-023-05365-9. PMID 37974160
- [Derived] McCaffrey J, Hunter A. Protocol Development for a Qualitative Methodological Study Within a Trial (Qual-SWAT): The KARMA-Dep-2 Trial. HRB Open Res. 2023 Nov 20;6:29. doi: 10.12688/hrbopenres.13721.2. eCollection 2023. PMID 37361338
- See also: Research Team Website — https://www.tcd.ie/medicine/psychiatry/research/depression-neurobiology-research-group/